CLINICAL TRIAL: NCT01917643
Title: A U.S. Retrospective Database Analysis Evaluating the Comparative Effectiveness of Budesonide/Formoterol (BFC) and Tiotropium Bromide Among COPD Patients
Brief Title: Comparative Effectiveness of Symbicort vs. Spiriva Among COPD Patients
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: HealthCore, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 000202; 000202 (Other: Astrazeneca)
Record Dates: First submitted 2013-07-31; First posted 2013-08-07 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: COPD Exacerbation
Keywords: COPD, Comparative Effectiveness, Symbicort
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Symbicort: BFC patients new to ICS/LABA and LAMA therapies
- Spiriva: Tiotropium bromide patients new to ICS/LABA and LAMA therapies

SUMMARY:
This study is intended to evaluate treatment effectiveness with budesonide/formoterol (BFC) and tiotropium tromide in patients new to ICS/LABA combination and LAMA therapies.

DETAILED DESCRIPTION:
Using US claims data from the HealthCore Integrated Research Environment, COPD patients ≥40 years old initiating BFC or tiotropium between 3/1/2009-2/28/2012 and considered at risk for a future exacerbation were identified and followed for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Continuous health plan enrollment for 12 months before and after index Rx
* At least one prescription fill for BFC or tiotropium bromide during intake period, and naive to ICS/LABA combination or LAMA therapies in year prior to first prescription claim.
* COPD diagnosis, and aged 40 years of age at time of first prescription
* At risk population for COPD exacerbations

Exclusion Criteria:

* ICS/LABA combination or LAMA therapy during pre-index period
* Patients with prescription claim for budesonide/formoterol and tiotropium bromide on the same day
* Patients diagnosed with cancer
* Patients with long-term OCS medication use during pre-index period

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Health plan members with COPD aged 40 years or older receiving one or more prescriptions of BFC or tiotropium bromide during 3/1/2009 and 1/31/2012 who are naive to ICS/LABA and LAMA combination therapies.
Sampling Method: Non-Probability Sample
Enrollment: 2396 (Actual)
Dates: Start 2013-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Time to first COPD exacerbation | 12 months
  The time to first COPD exacerbation will be calculated as the date of first COPD exacerbation minus index date. A COPD exacerbation event is defined as any of three conditions: COPD related inpatient hospitalization, COPD related emergency department visit, or COPD outpatient/office visit with a pharmacy claim for OCS and/or antibiotics on the same day or within ten days.

SECONDARY OUTCOMES:
COPD exacerbation rates | 12 months
  The rate of COPD exacerbation will be defined as the total number of COPD exacerbations during the post-index period for all patients in each treatment cohort divided by the total number of person years.
COPD respiratory medication use | 12 months
COPD related utilization | 12 months
  COPD related outpatient/office visit, COPD related inpatient hospitalization length of stay , COPD related ICU admission and length of stay, COPD procedures.
All-cause utilization | 12 months
  Frequency of all-cause resource use of: inpatient hospitalizations and length of stay, ICU admissions and length of stay, and outpatient/office visits. Total number of different prescription medication classes filled will also be determined.
All-cause and COPD related healthcare costs | 12 months
  Costs will be reported for the following resource uses: inpatient hospitalizations, ED visits, outpatient/office visits, skilled nursing facility, total medical, and prescriptions. Costs will be reported for all-cause as well as COPD related.
Treatment patterns and adherence | 12 months
  Continuity of care during the 12 month post-index period will be measured with the Bice and Boxerman index. Proportion of Days Covered (PDC) and Medication Possession Ration (MPR) will be used to measure the compliance of index medication (Symbicort or Spiriva) during the 12 month post-index period.
Treatment modification | 12 months
  COPD medication use, such as treatment changes, will be captured post-index.

REFERENCES:
- See also: Redacted protocol of Study 000202 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1870&filename=RedactedProtocolSymbicort_vs_SpirivaStudy000202.pdf
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1870&filename=NCT01917643_SYM_SPIRIVA_Redacted.pdf